CLINICAL TRIAL: NCT03292991
Title: REgistry of Selective Internal Radiation Therapy in TaiwaN (RESIN)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Collaborators: Kaohsiung Veterans General Hospital. (Other); National Taiwan University Hospital (Other); National Cheng-Kung University Hospital (Other); China Medical University Hospital (Other); Chang Gung Memorial Hospital (Other); Mackay Memorial Hospital (Other)
Responsible Party: Principal Investigator, vghtpe user, Principal Investigator, Dr. Rheun-Chuan Lee, Taipei Veterans General Hospital, Taiwan
Other Study IDs: QCR14021
Record Dates: First submitted 2017-08-04; First posted 2017-09-26 (Actual); Last update posted 2017-09-26 (Actual); Status verified 2017-09

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular Carcinoma; SIR Spheres; SIRT
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
All study objectives will be assessed in HCC patients or colorectal cancer patients with secondary metastases in the liver, respectively.

DETAILED DESCRIPTION:
All study objectives will be assessed in HCC patients or colorectal cancer patients with secondary metastases in the liver, respectively.

1. Primary objective:

   * To observe the safety of SIR-Spheres® microspheres therapy (SIRT)by,

     * Adverse events and serious adverse events (non-specific and radiation specific)
     * Changes in liver function parameters
   * To observe the efficacy of SIR-Spheres® microspheres therapy by, assessing the best overall response rate after SIRT
2. Secondary objectives:

   * To observe the efficacy of SIRT by,

     * Overall survival (OS)
     * Overall/objective response rate (ORR)
     * Time-to-progression
     * Time-to-liver progression
     * Progression-free survival
   * To observe the changes in clinical presentation after SIRT by,

     * ECOG score
     * Child-Pugh score
     * Percentage of subjects with down-staging or down-sizing of treated lesion to resection, transplantation, or radiofrequency ablation (RFA)
   * To observe the practice pattern of SIRT by,

     * Median dosage (GBq)
     * Number of SIRT sessions received by subjects
3. Exploratory objectives:

   * To explore prognostic factors for disease progression after SIRT by comparing the following parameters:

     * Number of tumors in subjects prior to SIRT
     * Median tumor size in subjects prior to SIRT
     * Location of tumor in subjects treated with SIRT (hepatic segment or lobe)
     * Number of prior TACE treatment in subjects
     * Antiviral therapy subjects HCC

ELIGIBILITY:
Inclusion Criteria, Patients who meet all inclusion criteria will be included:

* Males or non-pregnant females, at least 18 years of age (inclusive).
* Patients with clinically confirmed hepatocellular carcinoma (HCC) OR adenocarcinoma of colon/rectum with liver metastasis.
* Patients with liver dominant disease.
* Tumor burden ≤ 70% of total liver volume.
* HCC patients with child-Pugh Score class A or B.
* HCC patients with Barcelona-Clinic Liver Cancer (BCLC) stage A-C.
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0-1.
* Patients who are unsuitable for resection or immediate liver transplantation or who cannot be optimally treated with local ablation.
* Patients who have provided written informed consent.

Exclusion Criteria, Patients who meet any exclusion criteria will be excluded:

* Patients known to be hypersensitive to any component of study product.
* Female patients who are pregnant or lactating. Women of child bearing potential who disagree to practice medically recognized birth control methods throughout the study (from Screening to approximately 6 months post SIRT). Medically recognized birth control methods include hormonal contraceptives, intrauterine device/IUD, barrier device, or abstinence. With the exception of women who had been surgically sterilized (defined as having undergone hysterectomy or bilateral oophorectomy or bilateral salpingectomy; tubal ligation alone is not considered sufficient), or one year post-menopausal.

Withdrawal criteria:

* Patients consent withdrawal.
* Lost to follow-up for 2 consecutive visits.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HCC patients or colorectal cancer patients with secondary metastases in the liver.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2015-06-09 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Safety as per CTCAE 4.03, incidence of AEs and baseline change in liver function paired t-test or Wilcoxon signed rank test. | 6 months
  Toxicity will be accessed according to CTCAE v4.03. The incidence of adverse events will be summarized and the change in baseline liver function will be assessed by paired t-test or Wilcoxon signed rank test.

SECONDARY OUTCOMES:
Overall survival | 1 year
  Overall survival (OS) is determined for all enrolled subjects from Day 0 to the date of death or last contact.
Overall Response Rate per RECIST 1.1 and mRECIST | 1 year
  Liver tumor assessments for CRC will be evaluated by RECIST v1.1; and tumor assessments for HCC will be evaluated by mRECIST.
  - Objective Response Rate is defined as the proportion of subjects with tumor size reduction (i.e. the combined proportion of subjects with CR and PR) from Day 0 until documented tumor progression.
Time-to-progression per RECIST 1.1 and mRECIST | 1 year
  The time-to-progression (TTP) is calculated by the time from Day 0 to the date of disease progression (PD).
Time-to-liver progression per RECIST 1.1 and mRECIST | 1 year
  The time-to-liver progression is calculated by the time from Day 0 to the date of tumor progression (PD) in intrahepatic lesions.
Progression-free survival | 1 year
  Progression free survival (PFS) is determined for all enrolled patients from Day 0 until tumor progression or patient death.
Liver resection rate | 1 year
  Patients will be assessed for suitability for liver resection every study visit during the study period.
Liver transplantation rate | 1 year
  Patients will be assessed for suitability for liver transplantation every study visit during the study period.

CONTACTS AND LOCATIONS:
Overall Officials: Rheun-Chuan Lee, M.D., Principal Investigator — Taipei Veterans General Hospital, Taiwan
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan